CLINICAL TRIAL: NCT00978224
Title: Efficacy of Viusid Administration in Subjects With Chronic Inflammatory Syndrome Under Hemodialysis Treatment
Brief Title: Viusid Administration in Subjects With Chronic Inflammatory Syndrome Under Hemodialysis Treatment
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision of the investigator
Sponsor: Catalysis SL (Industry)
Responsible Party: Mirna Atiés Sánchez, Institute of Nephrology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0907-CU
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Inflammatory Syndrome
Keywords: dietary supplement; hemodialysis; Chronic Inflammatory Syndrome; Viusid
MeSH Terms: interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Viusid in combination with standard treatment for Chronic Inflammatory Syndrome including hemodialysis and the administration of a hypercaloric and hyperproteic diet
  Interventions: Dietary Supplement: Viusid
- B (Placebo Comparator): Placebo in combination with standard treatment for Chronic Inflammatory Syndrome including hemodialysis and the administration of a hypercaloric and hyperproteic diet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Viusid — 3 Viusid bags (Orally administered) per day, for 60 weeks
  Arms: A
Dietary Supplement: Placebo — 3 Placebo bags (Orally administered) per day, for 60 weeks.
  Arms: B

SUMMARY:
The purpose of the study is to determine whether Viusid administration improves malnutrition, atherosclerosis, erythropoietin response and the frequency of infection episodes in subjects with Chronic Inflammatory Syndrome under hemodialysis treatment. The duration of this double-blind placebo controlled phase 3 clinical trial will be 60 weeks. All patients enrolled in the study will be receiving the standard treatment for Chronic Inflammatory Syndrome including hemodialysis and administration of a hypercaloric and hyperproteic diet. Efficacy assessment will be carried out 12 weeks after the end of Viusid or placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic terminal nephropathy under hemodialysis treatment for at least 3 months
* Signed informed consent

Exclusion Criteria:

* Patients with chronic terminal nephropathy previously treated with peritoneal dialysis
* Receptors of a renal graft
* Patients with malignant neoplastic conditions
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) at week 72 (end of the treatment) | 72 weeks
Carotidal Doppler at week 72 (end of the treatment) | 72 weeks
C reactive protein at weeks 72 (end of the treatment) | 72 weeks
Hemoglobin at week 72 (end of the treatment) | 72 weeks

SECONDARY OUTCOMES:
Cholesterol at week 72 | 72 weeks
Triglycerides at week 72 | 72 weeks
Frequency of infection episodes at week 72 | 72 weeks
Creatinine at week 72 | 72 weeks
Uric acid at week 72 | 72 weeks
Glutamic-pyruvic transaminase (GPT)at week 72 | 72 weeks
Glutamic-oxaloacetic transaminase (GOT)at week 72 | 72 weeks
Blood glucose concentrations at week 72 | 72 weeks
Gasometry at week 72 | 72 weeks
Adverse effects at week 72 | 72 weeks
Albumin at week 72 | 72 weeks
KTV at week 72 | 72 weeks
Phosphocalcic metabolism at week 72 | 72 weeks
Hematocrit at week 72 | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mirna Atiés Sánchez, MD, Principal Investigator — Institute of Nephrology "Dr. Abelardo Buch López"
Locations (1):
- Institute of Nephrology "Dr. Abelardo Buch López", Havana, Cuba